CLINICAL TRIAL: NCT00083083
Title: Positron Emission Tomography Pre- and Post-treatment Assessment For Locally Advanced Non-Small Cell Lung Carcinoma
Brief Title: Fludeoxyglucose F18 Positron Emission Tomography Imaging In Assessing Patients Before and After Treatment for Locally Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Radiation Therapy Oncology Group (Network)
Responsible Party: Mitchell Machtay, Kimmel Cancer Center at Thomas Jefferson University - Philadelphia
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000362061; ACRIN-6668; RTOG-0235; NCT00194389 (obsolete NCT alias)
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2007-10

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Cisplatin; Docetaxel; Etoposide; Paclitaxel; Vinblastine; Vinorelbine; Gene Expression Profiling; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: docetaxel
Drug: etoposide
Drug: paclitaxel
Drug: vinblastine sulfate
Drug: vinorelbine tartrate
Genetic: gene expression analysis
Procedure: positron emission tomography
Radiation: fludeoxyglucose F 18
Radiation: radiation therapy

SUMMARY:
RATIONALE: Imaging procedures, such as fludeoxyglucose F18 positron emission tomography (^18FDG-PET), may improve the ability to detect disease progression and help doctors predict a patient's response to treatment and plan more effective treatment.

PURPOSE: This phase II trial is studying how well ^18FDG-PET imaging works in detecting disease progression and determining response to treatment in patients who are undergoing chemoradiotherapy for locally advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether peak standardized uptake value (SUV) for fludeoxyglucose F 18 positron emission tomography (FDG-PET) shortly after definitive chemoradiotherapy is predictive of long-term survival of patients with inoperable stage IIB or III non-small cell lung cancer.

Secondary

* Determine whether max SUV for FDG-PET shortly after definitive chemoradiotherapy is predictive of long-term survival in these patients.
* Determine whether post-treatment imaging using peak and max SUV for FDG-PET shortly after definitive chemoradiotherapy is predictive of local disease control in these patients.
* Determine whether pre-treatment imaging using these techniques is predictive of long-term survival and local disease control in these patients.
* Correlate, if possible, Ki-67 expression with overall survival of patients assessed with these imaging techniques.

OUTLINE: This is a diagnostic, multicenter study.

Before starting chemoradiotherapy, patients undergo baseline whole-body positron emission tomography (PET) imaging. Patients receive fludeoxyglucose F 18 (^18FDG) IV followed 50-70 minutes later by PET imaging. Patients then receive concurrent definitive radiotherapy and chemotherapy. Patients enrolled in other treatment-oriented clinical trials receive therapy as per that trial. Other patients receive standard thoracic radiotherapy (dose ≥ 60 Gy) and standard chemotherapy comprising a platin (cisplatin or carboplatin) and a second non-platin, non-gemcitabine drug (etoposide, vinblastine, vinorelbine, paclitaxel, or docetaxel). Approximately 14 weeks after completion of chemoradiotherapy and adjuvant chemotherapy (if given), patients undergo post-treatment ^18FDG-PET imaging.

Patients are followed every 3 months for 2 years and then every 6 months for at least 1 year.

PROJECTED ACCRUAL: A total of 250 patients (including at least 75 with stage IIB/IIIA disease and at least 75 with stage IIIB disease) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC)

  * Clinical stage IIB or III disease
  * No small cell carcinoma
  * No stage IV disease*
  * No diffuse bronchoalveolar subtype
  * No planned definitive surgical resection NOTE: *Patients with evidence of stage IV disease by positron emission tomography are eligible if the evidence cannot be confirmed by other means AND the physician still plans to proceed with definitive chemoradiation
* Planning treatment with definitive chemoradiotherapy

  * May be treated on another Radiation Therapy Oncology Group protocol (except phase I studies) OR with conventional concurrent NSCLC chemoradiotherapy
  * Radiotherapy ≥ 60 Gy AND chemotherapy to include concurrent platinum-based therapy
* No brain metastases by head CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Medically suitable for early concurrent chemoradiotherapy (radiotherapy dose ≥ 60 Gy)
* Able to tolerate positron emission tomography imaging
* No poorly controlled diabetes (defined as fasting glucose level > 200 mg/dL)
* No other malignancy within the past 3 years except basal cell or squamous cell skin cancer or carcinoma in situ
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No anticipated use of adjuvant biologic therapy beyond 14 weeks after the completion of radiotherapy

Chemotherapy

* See Disease Characteristics
* No anticipated use of adjuvant chemotherapy beyond 14 weeks after the completion of radiotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior thoracic radiotherapy
* No concurrent intensity-modulated radiotherapy

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2005-03; Primary Completion 2006-06 (Estimated)

PRIMARY OUTCOMES:
Relationship of survival to post-treatment peak standardized uptake value (SUV) as determined by the imaging institution

SECONDARY OUTCOMES:
Relationship of survival to post-treatment max SUV as determined by the imaging institute
Relationship of local control to post-treatment peak and max SUV as determined by the imaging institution
Relationship of survival and of local control to pre-treatment peak and max SUV as determined by the imaging institution
Reliability between peak and max SUV measurements both pre- and post-treatment
Proportion of participants who are either upstaged or downstaged by positron emission tomography scan
Reliability between PET scan-defined response to therapy measurements
Correlation of Ki-67 expression with peak and max pre-treatment SUV
Association between Ki-67 expression and overall survival at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Machtay, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (49):
- United States (46):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Scottsdale Medical Imaging, Limited, Scottsdale, Arizona
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Radiological Associates of Sacramento Medical Group at Sutter Cancer Center, Sacramento, California
  - Hospital of Saint Raphael, New Haven, Connecticut
  - Bethesda Comprehensive Cancer Care Center at Bethesda Memorial Hospital, Boynton Beach, Florida
  - North Broward Medical Center, Dearfield Beach, Florida
  - Integrated Community Oncology Network at Baptist Cancer Institute, Jacksonville, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Rush Cancer Institute at Rush University Medical Center, Chicago, Illinois
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber Partners Cancer Care, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Mallinckrodt Institute of Radiology at Washington University Medical Center, St Louis, Missouri
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Sister Patricia Lynch Regional Cancer Center at Holy Name Hospital, Teaneck, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Brown University School of Medicine, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Bon Secours Cancer Institute at St. Mary's Hospital, Richmond, Virginia
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
- Canada (2):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchner, Ontario
- National Cancer Center - Korea, Goyang, South Korea